CLINICAL TRIAL: NCT06729840
Title: Vitamin D in Keloids
Brief Title: Intralesional Treatment of Keloids
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sama Alaaeldin Ahmed, Sohag, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med--24-11-05MS
Record Dates: First submitted 2024-12-02; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Scar, Hypertrophic
Keywords: keloids , vitamin D
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid | interventions — Injections

STUDY DESIGN:
Intervention Model Description: 3 groups
Who Masked: Participant
Masking Description: Participant doesnot know injected substance
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Will include 15 patients will injected with vitamin D
  Interventions: Drug: Injection
- Group 2 (Active Comparator): Will include 15 patients will injected with botulinum toxin type A
  Interventions: Drug: Injection
- Group 3 (Active Comparator): Will include 15 patients will injected with triamcinolone acetonide
  Interventions: Drug: Injection

INTERVENTIONS:
Drug: Injection — Vitamin D , botox , tramcinolone intralesionally injected in keloid

SUMMARY:
Intralesional injection in treatment of keloid

DETAILED DESCRIPTION:
Our study will include 45 patient diveded into three groups , follow up will done before each session , 3month after the last session using photographing assessment , scoring , dermoscope

ELIGIBILITY:
Inclusion Criteria:

Both sex aged 18-60 having keloid

-

Exclusion Criteria:

* pregnancy , lactation Skin disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Posas score | One session every two weeks total duration 3 months
  patient and observer parameters will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No